CLINICAL TRIAL: NCT03804398
Title: Effect of Compliance Guided an Optimal Positive End-Expiratory Pressure on Arterial Oxygenation and Intrapulmonary Shunt During One-lung Ventilation
Brief Title: Effect of Optimal Positive End-Expiratory Pressure on Oxygenation and Intrapulmonary Shunt During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FujianUnionAnethesiaOne
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimal PEEP group (Experimental): The study group titrate PEEP from 4cmH2O,increased in 2cmH2O steps and hold at each step for 1min,and the static pulmonary compliance(Cst) would be record.Optimal PEEP was determined until the maximal static pulmonary compliance was obtained
  Interventions: Device: compliance guided an optimal Positive End-Expiratory Pressure
- PEEP level of 5 cmH2O group (Active Comparator): In the control group at PEEP level of 5 cmH2O was established and maintained during the study period
  Interventions: Device: PEEP level of 5 cmH2O

INTERVENTIONS:
Device: compliance guided an optimal Positive End-Expiratory Pressure — The study groups received an alveolar recruitment maneuver(increase inspiratory pressure to 30cmH2O for 10s) at the 10min after one-lung ventilation. After the alveolar recruitment maneuver,the study group titrate PEEP from 4cmH2O,increased in 2cmH2O steps and hold at each step for 1min,and the static pulmonary compliance(Cst) would be record.Optimal PEEP was determined until the maximal static pulmonary compliance was obtained.
  Arms: optimal PEEP group
Device: PEEP level of 5 cmH2O — In the control group at PEEP level of 5 cmH2O was established and maintained during the study period
  Arms: PEEP level of 5 cmH2O group

SUMMARY:
To observe the effect of compliance guided an optimal Positive End-Expiratory Pressure（PEEP）on arterial oxygenation and intrapulmonary shunt during one-lung ventilation(OLV)，and discuss the lung protective effect of optimal PEEP during one-lung ventilation.

DETAILED DESCRIPTION:
Sixty patients undergoing thoracic surgery were randomly allocated to the study or control group.Patients were monitored for electrocardiogram, pulse oximetry, and non-invasive blood pressure,20 gauge cannula needle for radial artery catheterization under local anesthesia, monitoring ABP.,the right subclavian vein was selected for catheterization under local anesthesia,monitoring CVP.Anesthesia was induced with sufentanil 0.4 μg/kg, propofol 2 mg/kg, and cisatracurium 0.3 mg/kg.The trachea was intubated with a double-lumen tube (DLT)，37F for male and 35F for female patients.Tube position was confirmed by bronchoscopy in the supine and lateral positions.Anesthesia was maintained with sevoﬂurane 1.0-1.5 vol%，propofol 2-4 mg/(kg·h) and remifentanil 0.1-0.2 μg/(kg·min) and intermittent cisatracurium 0.06-0.1 mg/kg.The lungs were initially ventilated using a volume-controlled ventilation mode,two-lung ventilation(TLV):tidal volume (VT) 8 ml/kg,respiratory rate 12-14 bpm, inspiratory:expiratory (I:E) ratio 1:2, in 60% oxygen without PEEP. During OLV, VT was reduced to 6 ml/kg,OLV was initiated at the moment of skin incision.Both groups received an alveolar recruitment maneuver(increase inspiratory pressure to 30cmH2O for 10s) at the 10min after one-lung ventilation. After the alveolar recruitment maneuver,the study group titrate PEEP from 4cmH2O,increased in 2cmH2O steps and hold at each step for 1min,and the static pulmonary compliance(Cst) would be record.Optimal PEEP was determined until the maximal static pulmonary compliance was obtained.In the control group at PEEP level of 5 cmH2O was established and maintained during the study period.Blood gas analyses, respiratory variables, and hemodynamic variables were recorded at 6 different time points:10 min after TLV(T0), 10min after OLV(T1), 30min after PEEP(T2), 60min after PEEP(T3), 10min after the end OLV(T4) and 20min after extubation(T5).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 yr to 65 yr
* Body mass index(BMI)18-28kg/m2
* American Society of Anesthesiologists Physical Status Classifications I to II
* Normal cardiac and pulmonary function
* Diagnosed with uncomplicated lung cancer and was to receive video-assist thoracoscopic lobectomy under general anesthesia.

Exclusion Criteria:

* Forced expiratory volume at one second/forced vital capacity <70%
* Asthma
* Chronic obstructive pulmonary disease
* Acute lung infection
* Past history of thoracic surgery
* Cardiac,hepatic,renal and endocrine diseases
* Preoperative glucocorticoid medication
* Preoperative chemotherapy
* Peripheral oxygen saturation（SpO2） kept below 90% for more than 10 minutes during operation
* Blood transfusion during operation
* Duration of one-lung ventilation less than an hour
* Occurrence of severe complications like allergic shock

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
arterial oxygenation | 24 hours
  To observe the effect of compliance guided an optimal Positive End-Expiratory Pressure（PEEP）on arterial oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua chen, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- FujianUnionHospital, Fuzhou, Fujian, China